CLINICAL TRIAL: NCT02236234
Title: Immune Response to HPV Vaccine Among HIV-1-infected Subjects in Brazil
Acronym: HPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jorge Casseb, PI, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010/07076-4; FAPESP (Other Grant/Funding Number: 2010/07076-4)
Record Dates: First submitted 2014-04-17; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Infection
Keywords: HIV; HPV; Clinical trial; outcome
MeSH Terms: conditions — Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Experimental): one group with HPV vaccine
  Interventions: Biological: HPV vaccine

INTERVENTIONS:
Biological: HPV vaccine — HPV vaccine
  Other Names: cerverix

SUMMARY:
Besides the specific response to vaccine antigens, the investigators will analyze the anti-HPV immune response in HIV-1-infected men in different strata of immune deficiency. The hypothesis will be tested by stratification by T CD4 + lymphocytes in an attempt to assess the range of the count with the highest possibility of vaccine response. Thus, knowledge of vaccine response in HIV-infected patients, indicate which patients would have greater potential for vaccine response in vivo.

DETAILED DESCRIPTION:
The study will be divided into three groups. Patients with HIV-1 infection will be subdivided into groups according to T CD4 + lymphocytes at the time of vaccination: Over 500 CD4 T cells count and bellow 500 CD4 T cells count. A healthy control group will be also studied.

ELIGIBILITY:
Inclusion Criteria: HIV

* Men with age between 35 and 45 years of age.

Exclusion Criteria:

* Current or previous infection with human papillomavirus (HPV)

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Presence of Anti-HPV antibody titers | 0, 30 and 180 days of vaccination anti-HPV
  The anti-HPV titers will be compared from baseline to the date of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: jorge casseb, phD, Principal Investigator — USP
Locations (1):
- Institute of Tropical Medicine of Sao Paulo, São Paulo, São Paulo, Brazil